CLINICAL TRIAL: NCT01803724
Title: Comparison Between Lactulose and Glucose Breath Tests as Predictors of Clinical Benefit From Rifaximin in Irritable Bowel Syndrome Patients
Brief Title: Lactulose and Glucose Breath Tests as Predictors of Clinical Benefit From Rifaximin in Irritable Bowel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: PUC-0003
Record Dates: First submitted 2013-03-01; First posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Small Intestinal Bacterial Overgrowth; Lactulose breath test; Glucose breath test; Rifaximin
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Irritable Bowel Syndrome (IBS) is a frequent disease, affecting between 10 and 20% of general population. Several pathophysiologic mechanisms have been described in IBS, among them the role of intestinal microbiota and small intestinal bacterial overgrowth (SIBO) have received special attention. SIBO has an adequate response to antibiotic treatment, unfortunately it didn't have an adequate diagnostic test: The classic gold standard -jejunal aspirate culture- has been criticized due to lack of standardization; the breath tests are simpler and widely available, but they have also been criticized due to inadequate diagnostic accuracy for SIBO. For this reason seems important to evaluate the performance of breath tests in terms of predicting clinical benefit of antibiotic therapy in IBS patients, rather than predicting a positive culture and SIBO.

The objectives of this study are:

1. Determine which breath test (lactulose or glucose) predicts better a potential clinical benefit of antibiotic treatment (Rifaximin) in IBS patients.
2. Determine which of the multiples diagnostic criteria described for the lactulose breath test predicts better a potential clinical benefit Rifaximin in IBS patients.

DETAILED DESCRIPTION:
After signing the informed consent, all patients will be submitted to both glucose and lactulose breath tests within a 10 days period. The order of the test will be randomized using a random number list of allocation, which will not be known by the patient. For the lactulose test a 10 g and for the glucose test a 50 g dose will be used, as previously suggested.

After the second test, patients will receive Rifaximin 400 mg TID (1200 mg/day) for 10 days. In the case of methane producers (defined as patients with basal methane levels > 3 ppm) Neomycin 500 mg BID (1000 mg/day) for ten days will be added, as suggested by Low et al.

Two weeks after the antibiotic course, patients will be cited and the following data will be assessed: 1. Adequate relief for global IBS symptoms. 2. Adequate relief for bloating. 3. Evaluation of IBS severity using IBSSS. 4. Drug induced side effects. Only after that information is submitted by the patient, the results of the test will be revealed.

Patients will be classified as responders or not according to their global symptoms adequate relief status. Using this as gold standard criterion, the test performance, in terms of sensitivity, specificity, positive and negative predictive value, will be calculated for the following tests:

1. Glucose breath test. A ROC curve will be calculated to determine the best cutoff value
2. Lactulose breath test using the rise occurring before 60 min, without the presence of a double peak. A ROC curve will be calculated to determine the best cutoff value
3. Lactulose breath test using the rise occurring before 60 min, if there is a double peak. A ROC curve will be calculated to determine the best cutoff value
4. Lactulose breath test using the rise occurring before 90 min, without the presence of a double peak. A ROC curve will be calculated to determine the best cutoff value
5. Lactulose breath test using the rise occurring before 90 min, if there is a double peak. A ROC curve will be calculated to determine the best cutoff value

The different tests will be compared in terms of their performance at the optimal cutoff value and calculating the area under the ROC curve.

The sample size was calculated as previously suggested. Using Shah et al data, we assumed a sensitivity of 72% and a specificity of 66% for the lactulose breath test. Using an alpha and beta error of 5% and 20%, respectively, and a disease prevalence of 35% (SIBO in IBS), we estimate a sample size of 120 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting Rome III criteria for IBS.

Exclusion Criteria:

1. Patients < 18 years old
2. Previous intestinal (small or large bowel) resection
3. Known anatomical intestinal alterations, including diverticula and stenosis
4. Inflamatory bowel disease (Crohn´s or ulcerative colitis)
5. Presence of IBS alarm signs suggestive of organic disease, including anemia or family history of celiac disease or colon cancer
6. Recent acute onset diarrhea
7. Pregnancy
8. Neurologic or psychiatric disease that may not allow the patient to appropriately describe clinical outcomes
9. Presence of a disease that could affect intestinal transit, such as Parkinson´s, Chronic Intestinal Pseudobstruction, Scleroderma, Diabetes mellitus, etc
10. Impossibility to transitory withdraw drugs that affect intestinal transit, such as Calcium channel blockers, tricyclics
11. Inability to sign or rejection to informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting Rome III criteria for IBS.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Adequate relief for global IBS symptoms | Two weeks after the antibiotic course
  Adequate relief corresponds to the answer of the patient (yes or no) to the question ´have you achieved adequate relief from your symptoms?¨

SECONDARY OUTCOMES:
Evaluation of IBS severity using IBSSS | Two weeks after antibiotic course
  IBSSS is a score (mainly visual analogue scale (VAS) based) consisting of several questions regarding different IBS symptoms. The binary outcome adequate relief and a severity evaluation by IBSSS are the recommended outcomes by the designing of clinical trials Rome committee.
  All patients will be characterized in terms of basal IBS severity using IBSSS (before to course of 10 days of antibiotics).
Adequate relief for bloating. | Two weeks after the antibiotic course
  Adequate relief of bloating corresponds to the answer of the patient (yes or no) to the question ´have you achieved adequate relief from your bloating?¨.
Drug induced side effects. | Two weeks after antibiotic course

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cisternas, MD, Study Director — Pontificia Universidad Catolica de Chile; Roberto Candia, MD, Principal Investigator — Pontificia Universidad Catolica de Chile; Patricio Ibañez, MD, Principal Investigator — Pontificia Universidad Catolica de Chile; Juan Pablo Ortega, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Department of Gastroenterology, Pontificia Universidad Catolica de Chile, Santiago, Metropolitan, Chile

REFERENCES:
- [Background] Parkes GC, Brostoff J, Whelan K, Sanderson JD. Gastrointestinal microbiota in irritable bowel syndrome: their role in its pathogenesis and treatment. Am J Gastroenterol. 2008 Jun;103(6):1557-67. doi: 10.1111/j.1572-0241.2008.01869.x. Epub 2008 May 29. PMID 18513268
- [Background] Lin HC. Small intestinal bacterial overgrowth: a framework for understanding irritable bowel syndrome. JAMA. 2004 Aug 18;292(7):852-8. doi: 10.1001/jama.292.7.852. PMID 15316000
- [Background] DuPont AW, DuPont HL. The intestinal microbiota and chronic disorders of the gut. Nat Rev Gastroenterol Hepatol. 2011 Aug 16;8(9):523-31. doi: 10.1038/nrgastro.2011.133. PMID 21844910
- [Background] Gasbarrini A, Corazza GR, Gasbarrini G, Montalto M, Di Stefano M, Basilisco G, Parodi A, Usai-Satta P, Vernia P, Anania C, Astegiano M, Barbara G, Benini L, Bonazzi P, Capurso G, Certo M, Colecchia A, Cuoco L, Di Sario A, Festi D, Lauritano C, Miceli E, Nardone G, Perri F, Portincasa P, Risicato R, Sorge M, Tursi A; 1st Rome H2-Breath Testing Consensus Conference Working Group. Methodology and indications of H2-breath testing in gastrointestinal diseases: the Rome Consensus Conference. Aliment Pharmacol Ther. 2009 Mar 30;29 Suppl 1:1-49. doi: 10.1111/j.1365-2036.2009.03951.x. PMID 19344474
- [Background] Design of Treatment Trials Committee; Irvine EJ, Whitehead WE, Chey WD, Matsueda K, Shaw M, Talley NJ, Veldhuyzen van Zanten SJ. Design of treatment trials for functional gastrointestinal disorders. Gastroenterology. 2006 Apr;130(5):1538-51. doi: 10.1053/j.gastro.2005.11.058. PMID 16678567
- [Background] Fleiss, J.L., Statistical methods for rates and proportions. 2d ed. Wiley series in probability and mathematical statistics. 1981, New York: Wiley. xviii, 321 p
- [Background] Flahault A, Cadilhac M, Thomas G. Sample size calculation should be performed for design accuracy in diagnostic test studies. J Clin Epidemiol. 2005 Aug;58(8):859-62. doi: 10.1016/j.jclinepi.2004.12.009. PMID 16018921
- [Result] Saito YA, Schoenfeld P, Locke GR 3rd. The epidemiology of irritable bowel syndrome in North America: a systematic review. Am J Gastroenterol. 2002 Aug;97(8):1910-5. doi: 10.1111/j.1572-0241.2002.05913.x. PMID 12190153
- [Result] Gwee KA. Irritable bowel syndrome in developing countries--a disorder of civilization or colonization? Neurogastroenterol Motil. 2005 Jun;17(3):317-24. doi: 10.1111/j.1365-2982.2005.00627.x. PMID 15916618
- [Result] Yang J, Lee HR, Low K, Chatterjee S, Pimentel M. Rifaximin versus other antibiotics in the primary treatment and retreatment of bacterial overgrowth in IBS. Dig Dis Sci. 2008 Jan;53(1):169-74. doi: 10.1007/s10620-007-9839-8. Epub 2007 May 23. PMID 17520365
- [Result] Di Stefano M, Malservisi S, Veneto G, Ferrieri A, Corazza GR. Rifaximin versus chlortetracycline in the short-term treatment of small intestinal bacterial overgrowth. Aliment Pharmacol Ther. 2000 May;14(5):551-6. doi: 10.1046/j.1365-2036.2000.00751.x. PMID 10792117
- [Result] Lauritano EC, Gabrielli M, Scarpellini E, Ojetti V, Roccarina D, Villita A, Fiore E, Flore R, Santoliquido A, Tondi P, Gasbarrini G, Ghirlanda G, Gasbarrini A. Antibiotic therapy in small intestinal bacterial overgrowth: rifaximin versus metronidazole. Eur Rev Med Pharmacol Sci. 2009 Mar-Apr;13(2):111-6. PMID 19499846
- [Result] Khoshini R, Dai SC, Lezcano S, Pimentel M. A systematic review of diagnostic tests for small intestinal bacterial overgrowth. Dig Dis Sci. 2008 Jun;53(6):1443-54. doi: 10.1007/s10620-007-0065-1. PMID 17990113
- [Result] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Result] Shah ED, Basseri RJ, Chong K, Pimentel M. Abnormal breath testing in IBS: a meta-analysis. Dig Dis Sci. 2010 Sep;55(9):2441-9. doi: 10.1007/s10620-010-1276-4. Epub 2010 May 14. PMID 20467896